CLINICAL TRIAL: NCT06325657
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLINDED, PLACEBO-CONTROLLED TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE IN PREGNANT PARTICIPANTS LIVING WITH HIV AND THEIR INFANTS
Brief Title: A Study to Learn About the Vaccine RSVpreF In Pregnant Participants With HIV and Their Infants
Acronym: MORISOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671032
Record Dates: First submitted 2024-03-08; First posted 2024-03-22 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory Tract Infection; HIV; Maternal; Vaccine
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSVpreF vaccine (Experimental): RSV vaccine (RSVpreF)
  Interventions: Biological: RSVpreF vaccine
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebp

INTERVENTIONS:
Biological: RSVpreF vaccine — RSVpreF vaccine
  Arms: RSVpreF vaccine
Biological: Placebp — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn about the safety and immune activity of the RSVpreF vaccine. It will be studied in infants born to mothers living with HIV. These infants may have higher chances of getting sick or dying due to RSV infection. Respiratory Syncytial Virus (RSV) is a common type of virus (germ) that can cause severe illness (airway diseases), where medical help is needed. Vaccines help your body make antibodies which help fight against diseases. The antibodies are substances your body uses to fight off an infection. The antibodies can be passed to the infant through the placenta of the mother.

The study will look at the safety, tolerability, and immune activity in mothers and their infants.

This study is seeking pregnant women who are:

* Less than or equal to 49 years old and have HIV (Human immunodeficiency virus -
* Receiving standard medical care during the pregnancy
* Do not have syphilis (bacterial sexually transmitted disease), Hepatitis B Virus ((HBV) liver infection), Tuberculosis ((TB) bacterial lung infection).
* Have been on stable (anti-retroviral) HIV treatment for more than or equal to 90 days.
* agree to be present for all study visits, procedures, and blood draws.

Participants will either receive:

* RSVpreF vaccine
* A placebo. A placebo does not have any medicine it but looks just like the study vaccine.

Pregnant participants will be involved in the study from:

* consent during their current pregnancy, and
* for 6 months after delivery of their baby (around 10 months in total). Pregnant participants will have at least 5 planned visits in this study. Infant participants: All eligible babies born to enrolled mothers will be followed up from birth for up to 6 months. Infant participants will have at least 3 study visits, with some site visits allowed to happen via home visits or over the telephone.

ELIGIBILITY:
Key Inclusion Criteria - Maternal Participants

* Women ≤49 years of age who are between 24 0/7 and 36 0/7 weeks of gestation on the day of planned vaccination, with an uncomplicated singleton pregnancy who are at no known increased risk for complications.
* Confirmed stable HIV disease.
* Current and stable use of antiretroviral therapy(ART) for at least 90 days prior to enrolment.
* Had a fetal anomaly ultrasound examination performed at ≥18 weeks of pregnancy with no significant fetal abnormalities observed.
* Intention to deliver at a hospital or birthing facility where study procedures can be obtained.
* Participant is willing to give informed consent for the participant's infant to participate in the study.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Key Inclusion Criteria - Infant Participants

* Evidence of a signed and dated ICD, signed by the parent(s)/legal guardian(s).
* Parent(s)/legal guardian(s) willing and able to comply with scheduled visits, investigational plan, laboratory tests, and other study procedures

Key Exclusion Criteria - Maternal Participants

* Prepregnancy body mass index (BMI) of >40 kg/m2 . If prepregnancy BMI is not available, the BMI at the time of the first obstetric visit during the current pregnancy may be used.
* Participant with opportunistic infections or malignancy.
* History of active chronic viral hepatitis with biochemical evidence of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values >5 times the upper limit of normal within 6 months before enrollment.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention or any related vaccine.
* Current pregnancy resulting from in vitro fertilization. Participants known to have used clomiphene citrate and/or letrozole with or without intrauterine insemination (IUI) are permitted.
* Current pregnancy complications or abnormalities at the time of consent that will increase the risk associated with the participation in and completion of the study, including but not l limited to the following:
* Preeclampsia, eclampsia, or uncontrolled gestational hypertension.
* Placental abnormality.
* Polyhydramnios or oligohydramnios.
* Significant bleeding or blood clotting disorder.
* Endocrine disorders, including untreated hyperthyroidism or untreated hypothyroidism. This also includes disorders of glucose intolerance (eg, diabetes mellitus type 1 or 2) antedating pregnancy or occurring during pregnancy if uncontrolled at the time of consent.
* Any signs of premature labor with the current pregnancy or having ongoing intervention (medical/surgical) in the current pregnancy to prevent preterm birth.
* Prior pregnancy complications or abnormalities at the time of consent, based on the investigator's judgment, that will increase the risk associated with the participation in and completion of the study, including but not limited to the following:
* Prior preterm delivery at ≤34 weeks' gestation
* Prior stillbirth or neonatal death
* Previous infant with a known genetic disorder or significant congenital anomaly
* Non-HIV-associated congenital or acquired immunodeficiency disorder, or rheumatologic disorder or other illness requiring chronic treatment with known immunosuppressant medications.
* Antituberculosis treatment use currently or at any time during this current pregnancy.

Key Exclusion Criteria - Infant Participants

• Infant who is a direct descendant (eg, child or grandchild) of the investigator site staff or sponsor and sponsor delegate employees directly involved in the conduct of the study.

Ages: 0 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 648 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Maternal Participants Primary Safety - The proportion of participants reporting systemic reactions | Within 7 days following study administration intervention
  Systemic Reactions: fever, fatigue, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded based on e-diary and participant reported reactogenicity events.
Maternal Participants Primary Safety - The proportion of participants reporting local reactions | Within 7 days following study administration intervention
  Local reactions included pain at injection site, redness and swelling recorded based on e-diary and participant reported reactogenicity events.
Maternal Participants Primary Safety - The proportion of participants reporting Adverse Events (AEs) | Through 1 month following study administration intervention
  An adverse event was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Adverse events included both serious and non-serious adverse events.
Maternal Participants Primary Safety - The proportion of participants reporting Adverse Event of Special Interests (AESIs) | Throughout the study duration (approximately 10 months)
  AESIs include preterm delivery, diagnosis of GB syndrome, Diagnosis of Acute polyneuropathy without underlying etiology, hypertensive disorders of pregnancy, atrial fibrillation.
Maternal Participants Primary Safety - The proportion of participants reporting Serious Adverse Events (SAEs) | Throughout the study duration (approximately 10 months)
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Infant Participants Primary Safety - The proportion of participants reporting Specific Birth Outcomes | Birth
  Describe specific birth outcomes for infant participants
Infant Participants Primary Safety - The proportion of participants reporting Adverse Events (AEs) | Through 1 month following birth
  An AE is any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs include both serious and non-serious adverse events.
Infant Participants Primary Safety - The proportion of participants reporting SAEs and Newly Diagnosed Chronic Medical Conditions (NDCMCs) | Throughout the study duration (approximately 6 months)
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
  NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects.

SECONDARY OUTCOMES:
Maternal Participants: Secondary Immunogenicity - GMT of NTs for RSV A and RSV B | Before vaccination and at the delivery visit
  GMT of NTs for RSV A and RSV B before vaccination and at the delivery visit
Maternal Participants: Secondary Immunogenicity - GMFR of NTs for RSV A and RSV B | From before vaccination and to the delivery visit
  GMFR of NTs for RSV A and RSV B from before vaccination to post vaccination blood-sampling visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- South Africa (14):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Josha Research, Bloemfontein, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - REIMED Reiger Park, Boksburg, Gauteng
  - Wits RHI, Johannesburg, Gauteng
  - University of Witwatersrand (WITS) - Vaccines and Infectious Diseases Analytics (VIDA), Johannesburg, Gauteng
  - Wits VIDA Nkanyezi Research Unit, Johannesburg, Gauteng
  - Setshaba Research Centre, Pretoria, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Qhakaza Mbokodo Research Clinic, Ladysmith, KwaZulu-Natal
  - Gole Biomed Research Centre, Polokwane, Limpopo
  - MRC Unit on Child And Adolescent Health, Cape Town, Western Cape
  - Gugulethu Green Clinic, Cape Town, Western Cape
  - FAMCRU - Worcester, Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Myer L, Wasserman E, Tabasum S, Shittu E, Liu Y, Jose L, Horne E, Moraba RS, Wilhase A, Zar HJ, Hussen N, Mogashoa MS, Malahleha M, Madhi SA, Sarwar UN, Snaggs H, Erdem R, Radley D, Kalinina EV, Pahud BA, Maddalena Lino M, Anastasiou OE, Swanson KA, Anderson AS, Gurtman A, Munjal I. Safety, Tolerability, and Immunogenicity of RSVpreF Vaccine in Pregnant Individuals Living with HIV. Vaccines (Basel). 2025 Dec 1;13(12):1218. doi: 10.3390/vaccines13121218. PMID 41441684
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671032